CLINICAL TRIAL: NCT01172106
Title: The Role of Psychoeducation on Perceived Social Support of Postpartum Others With a Psychotic Illness
Brief Title: Impact of Family Psychoeducation on Psychosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: Swedish International Development Cooperation Agency (SIDA) (Other Government)
Responsible Party: Janet Nakigudde, Department of Psychiatry, College of Health Sciences, Makerere University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2006/HD11/4572U
Record Dates: First submitted 2010-07-28; First posted 2010-07-29 (Estimated); Last update posted 2010-07-29 (Estimated); Status verified 2010-07

CONDITIONS: Postpartum Psychosis
Keywords: Postpartum psychosis; Perceived social support; Family psychoeducation
MeSH Terms: interventions — Psychosocial Intervention

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Encouragement on drug compliance (Placebo Comparator): The intervention for the placebo comparator will be encouragement on drug compliance
  Interventions: Behavioral: drug compliance; Behavioral: Encouragement of drug compliance
- Family psychoeducation (Experimental): The experimental group will receive weekly sessions of psychoeducation for 12 weeks in addition to receiving drug compliance encouragement
  Interventions: Behavioral: Family psychoeducation

INTERVENTIONS:
Behavioral: drug compliance — Mothers and their caregivers will be encouraged to comply with the given medication
  Other Names: Psychosocial intervention
  Arms: Encouragement on drug compliance
Behavioral: Encouragement of drug compliance — Mothers and their caregivers in the placebo comparator will receive an intervention of drug compliance encouragement
  Other Names: Psychosocial intervention
  Arms: Encouragement on drug compliance
Behavioral: Family psychoeducation — The experimental group will receive family psychoeducation for 12 sessions
  Other Names: Psychosocial intervention
  Arms: Family psychoeducation

SUMMARY:
There is currently no clear involvement of families/caregivers in the care for postpartum mothers that develop postpartum psychosis. The lack of knowledge on causes of postpartum psychosis may influence the nature of perceived social support that mothers receive from caregivers. It is hoped that the provision of a culturally adapted version of family psychoeducation will bridge the knowledge gap and provide the much needed information. We therefore hypothesized that the involvement of a family member of a postpartum mother with a psychotic illness in a weekly session of family psychoeducation.

DETAILED DESCRIPTION:
Postpartum psychosis causes distress to the mother, baby, spouse and other primary caregivers. This is especially true for Uganda where cultural beliefs for the causation of the illness place blame on supposedly the postpartum mother's promiscuity during pregnancy (COX, 1979). Cultural perceptions on the causes of postpartum psychosis may affect the nature of social support the mothers perceive from their families when they develop the illness. Other perceptions regarding postpartum psychosis in Uganda lay blame on supernatural causes like witchcraft.

Family psychoeducation which sets out to inform families of the nature of the illness is called for so as to demystify the illness.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum mothers with a psychiatric illness in the current postpartum period.
* Must have been admitted to the mental health facility for the current episode.

Exclusion Criteria:

* Mothers residing out of a radius of 50 km away from the health facility.
* Mothers that do not have caregivers.
* Mothers who are not fluent in the language in which the study will be conducted.

Ages: 13 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-09 (Estimated); Study Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
perceived social support of mothers | 3 months
  12 weekly sessions of family psychoeducation for a period of 3 months will improve perceived social support of mothers in the intervention arm.

SECONDARY OUTCOMES:
Improvement of psychological distress of the caregivers | 3 months
  12 weekly sessions of family psychoeducation with caregivers for a period of 3 months will improve psychological distress in caregivers of mothers that will have received family psychoeducation

CONTACTS AND LOCATIONS:
Overall Officials: Eija Airaksinen, Study Director — Karolinska Institutet
Locations (1):
- Makerere University College of Health Sciences, Kampala, Uganda